CLINICAL TRIAL: NCT01862315
Title: A Phase II Study of Hepatic Arterial Infusion (HAI) With Floxuridine (FUDR) and Dexamethasone (Dex) Combined With Systemic Gemcitabine and Oxaliplatin in Patients With Unresectable Intrahepatic Cholangiocarcinoma (ICC)
Brief Title: Hepatic Arterial Infusion (HAI) With Floxuridine (FUDR) and Dexamethasone (Dex) Combined With Systemic Gemcitabine and Oxaliplatin in Patients With Unresectable Intrahepatic Cholangiocarcinoma (ICC)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 13-066
Record Dates: First submitted 2013-05-20; First posted 2013-05-24 (Estimated); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Intrahepatic Cholangiocarcinoma; Peripheral Cholangiocarcinoma; Cholangiolar Carcinoma; Cholangiocellular Carcinoma
Keywords: Hepatic Arterial Infusion (HAI); Floxuridine (FUDR); Dexamethasone (DEX); Gemcitabine; Oxaliplatin; 13-066
MeSH Terms: conditions — Cholangiocarcinoma | interventions — Floxuridine; Dexamethasone; Gemcitabine; Oxaliplatin

ARMS (3):
- No prior chemo or responded/stable with prior chemo (Experimental): All patients receive HAI FUDR ([0.12 mg/kg/day kg 30] / pump flow rate)& dexamethasone ({1 mg/m2/day30} pump flow rate) on Day 1 of each cycle. Chemotherapy with HAI FUDR/Dex will commence no sooner than 14 days postsurgical placement of HAI pump. All patients receive Gemcitabine (800 mg/m2 IV over 30 minutes) & Oxaliplatin (85 mg/m2 IV over 120 minutes) on Days 1 & 15 of each cycle, however initiation with systemic chemotherapy will not take place until 4 weeks post-surgery for pump placement, so the first doses of systemic chemotherapy will be given on Cycle 1, Day 15, & then every 2 weeks thereafter. Clinical MRI examinations of the abdomen & pelvis are obtained at baseline following surgery, prior to treatment initiation & 4 weeks after initiation of HAI FUDR. Subsequently, the patient will undergo MRI approximately at months 3, 6 & 9 thereafter A non-contrast CT of chest, abdomen & pelvis will also be obtained as part of routine clinical care.
  Interventions: Drug: Floxuridine (FUDR); Drug: dexamethasone; Drug: Gemcitabine; Drug: Oxaliplatin; Other: MRI; Other: Research blood draws
- patients who have failed systemic therapy (Experimental): All patients receive HAI FUDR ([0.12 mg/kg/day kg 30] / pump flow rate)& dexamethasone ({1 mg/m2/day 30}/ pump flow rate) on day 1 of each cycle. Chemotherapy with HAI FUDR/Dex will commence no sooner than 14 days postsurgical placement of HAI pump. All patients receive Gemcitabine (800 mg/m2 IV over 30 minutes) & Oxaliplatin (85 mg/m2 IV over 120 minutes) on Days 1 & 15 of each cycle, however initiation with systemic chemotherapy will not take place until 4 weeks post-surgery for pump placement, so the first doses of systemic chemotherapy will be given on Cycle 1, Day 15, & then every 2 weeks thereafter. Clinical MRI examinations of the abdomen & pelvis are obtained at baseline following surgery, prior to treatment initiation & 4 weeks after initiation of HAI FUDR. Subsequently, the patient will undergo MRI approximately at months 3, 6 & 9 thereafter A non-contrast CT of chest, abdomen & pelvis will also be obtained as part of routine clinical care.
  Interventions: Drug: Floxuridine (FUDR); Drug: dexamethasone; Drug: Gemcitabine; Drug: Oxaliplatin; Other: MRI; Other: Research blood draws
- pts who have had prior oxaliplatin & have existing neuropathy (Experimental): All patients receive will receive gemcitabine alone with HAI FUDR/Dex Gemcitabine (800 mg/m2 IV over 30 minutes) alone on Days 1 and 15 of each cycle, however initiation with systemic chemotherapy will not take place until 4 weeks post-surgery for pump placement, so the first doses of systemic chemotherapy will be given on Cycle 1, Day 15, and then every 2 weeks thereafter.
  Interventions: Drug: dexamethasone; Drug: Gemcitabine; Other: MRI; Other: Research blood draws

INTERVENTIONS:
Drug: Floxuridine (FUDR)
  Arms: No prior chemo or responded/stable with prior chemo; patients who have failed systemic therapy
Drug: dexamethasone
Drug: Gemcitabine
Drug: Oxaliplatin
  Arms: No prior chemo or responded/stable with prior chemo; patients who have failed systemic therapy
Other: MRI
Other: Research blood draws — These are optional

SUMMARY:
The purpose of this study is to use both, liver pump treatment and systemic chemotherapy, to assess the effects this type of treatment has on the patient and the tumor. Liver pump treatment uses a metal pump that is surgically placed in the abdomen and gives chemotherapy directly to the liver. Systemic chemotherapy gives chemotherapy through a vein [intravenously (IV)] and treats the whole body. This type of treatment has been done before and had shown that people with both pump and systemic chemotherapy had improved results. The investigators hope that this combination of treatments improves the response to chemotherapy and reduces the spread of the disease.

Another purpose of this study is to learn the clinical importance of a specific type of MRI scan. The investigators would like to see if this type of MRI will help predict the response to the treatment and see if they could help the physician with their treatment plan. These scans will be done at specific time points.

The last purpose of this study is to learn more about how the tumor interacts with the chemotherapy. This will be done through a biopsy taken during surgery and blood draws at specific time points.

Permission from patients entering the study will be obtained to take normal and tumor liver biopsies at the time of surgery. These samples are voluntary and optional.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 21 years
* Histologically confirmed intrahepatic cholangiocarcinoma (also variously reported as peripheral cholangiocarcinoma, cholangiolar carcinoma or cholangiocellular carcinoma) (ICC). Confirmation of the diagnosis at MSKCC or at the enrolling institution must be obtained prior to initiation of protocol therapy.
* Clinical or radiographic evidence of metastatic disease to regional lymph nodes will be allowed, provided it is amenable to resection.
* Radiographically measurable disease. Measurable disease is defined as disease that can be assessed with 2-dimensional measurements on a cross-sectional imaging. Minimum lesion size is 2cm in greatest diameter as per RECIST criteria.
* Disease must be considered unresectable at the time of preoperative evaluation.
* Presence of less than 70% liver involvement by cancer.
* Patients may have failed ablative therapy
* Patient previously treated with systemic chemotherapy will be eligible
* KPS ≥ 60% and be considered candidates for general anesthesia, abdominal exploration and hepatic artery pump placement
* Patients with chronic hepatitis and/or cirrhosis are eligible, but must be Child-Pugh class A
* Patients must be able to read, understand and sign informed consent
* WBC ≥ 2,000 cells/mm3
* Platelet count ≥ 75,000/mm3
* Creatinine ≤ 1.8 mg/dl
* Total bilirubin < 1.5 mg/dl

Exclusion Criteria:

* Presence of distant metastatic disease. Patients will undergo radiographic evaluation to exclude the possibility of distant metastatic disease. For patients who have undergone pre- or postoperative biopsies that definitively diagnose ICC, the diagnostic studies may be modified at the discretion of the MSKCC Principal Investigator. Clinical or radiographic evidence of metastatic disease to regional lymph nodes will be allowed, provided it is amenable to resection.
* Prior treatment with FUDR
* Prior external beam radiation therapy to the liver
* Diagnosis of sclerosing cholangitis
* Clinical evidence or portal hypertension (ascites, gastroesophageal varices, or portal vein thrombosis) surgically related ascites does not exclude the patient)
* Active infection
* Pregnant or lactating women
* History of other malignancy within the past 3 years (except non-melanoma skin cancer)
* Life expectancy less than 12 weeks
* Inability to comply with study and/or followup procedures
* History of peripheral neuropathy (Note: this does not apply to Cohort 3)

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2013-05; Primary Completion 2025-03-18 (Actual); Study Completion 2025-03-18 (Actual)

PRIMARY OUTCOMES:
progression free survival for Cohort 1 | 6 months
  Treatment evaluation will be done using RECIST (version 1.1)
progression free survival for Cohort 2 | 3 months
  Treatment evaluation will be done using RECIST (version 1.1)
response for Cohort 3 | 6 months
  Treatment evaluation will be done using RECIST (version 1.1)

SECONDARY OUTCOMES:
Correlative objective of of dynamic contrast enhanced (DCE)-MRI imaging of intrahepatic cholangiocarcinoma before treatment and early during the course of treatment. | 1 year
  This study will investigate DCE-MRI as potential imaging biomarkers and will measure tumor perfusion parameters and diffusion coefficients before initiating treatment and on follow-up MRI scans during treatment.
Correlative objective of of dynamic contrast enhanced DWI of intrahepatic cholangiocarcinoma before treatment and early during the course of treatment. | 1 year
  This study will investigate diffusion weighted imaging (DWI) as potential imaging biomarkers and will measure tumor perfusion parameters and diffusion coefficients before initiating treatment and on follow-up MRI scans during treatment.

CONTACTS AND LOCATIONS:
Overall Officials: William Jarnagin, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (6):
- United States (6):
  - Memorial Sloan Kettering Cancer Center, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Commack, Commack, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Nassau, Uniondale, New York

REFERENCES:
- See also: Memorial Sloan-Kettering Cancer Center — http://www.mskcc.org/